CLINICAL TRIAL: NCT01038297
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND, WITHIN-SUBJECT CONTROLLED, DOSE-RANGING STUDY TO EVALUATE EFFICACY AND SAFETY OF EXC 001 FOR THE TREATMENT OF INCISION SCARS IN THE PANNUS OF SUBJECTS UNDERGOING AN ELECTIVE ABDOMINOPLASTY
Brief Title: Safety and Efficacy Study of Different Dose Levels of EXC 001 to Improve the Appearance of Scars in Subjects Undergoing Elective Abdominoplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXC 001-201; B5301009 (Other: Alias Study Number)
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Scar Prevention
Keywords: Scarring
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EXC 001 (Experimental)
  Interventions: Drug: EXC 001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EXC 001 — Intradermal injections of EXC 001 and placebo given on various schedules.
  Arms: EXC 001
Drug: Placebo — Intradermal injections of EXC 001 and placebo given on various schedules.
  Arms: Placebo

SUMMARY:
This study will compare how well EXC 001 works versus placebo in reducing the appearance of scars in subjects undergoing elective abdominoplasty. The study will also evaluate the safety of EXC 001 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have sufficient excess abdominal tissue to qualify for a standard elective abdominoplasty
* Subject has chosen to have an elective abdominoplasty
* Medically healthy with normal screening results
* Subjects must not be pregnant or lactating

Exclusion Criteria:

* Subjects with existing scars or significant striae on the abdominal pannus
* Females who are currently pregnant or pregnant during the 12 months prior to inclusion in the study, or lactating
* Participation in another clinical trial within 30 days prior to the start of the study
* Any other condition or prior therapy, which, in the opinion of the PI, would make the subject unsuitable for this study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2009-12-01 (Actual); Primary Completion 2010-07-07 (Actual); Study Completion 2010-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Northwestern University,Division of Plastic Surgery, Chicago, Illinois
  - Body Aesthetic Plastic Surgery, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=EXC001-201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had chosen and qualified (had sufficient excess abdominal tissue) for a standard elective abdominoplasty were recruited in this study. The study was conducted in two-parts: Part A (Skin Testing Phase) and Part B (Active Dosing Phase). Participants with negative skin sensitization in Part A entered into Part B .
Pre-assignment Details: Part B (incision wounds [IW] and abdominoplasty surgery): On Day 1, participants received 20 incisions (2 centimeters [cm] each), 10 incisions on either side of the midline (4 vertical columns of 4 incisions each, 2 columns of 2 incisions [lateral biomarker incisions]), on the abdominal area to be removed during abdominoplasty.
Groups:
- Cohort 1: EXC 001 and Placebo: In Part A participants received single intradermal injections of EXC-001 at a dose of 5 milligram (mg) on Day 1 and 21. Third 5 mg intradermal injection was administered at the discretion of Investigator based on the event of an equivocal skin sensitization on Day 38 or at least 7 days prior to surgery (Day 1 in Part B). The injection site was evaluated immediately after the injection and on Days 21, 28, 38, 50 until day of surgery. Participants with negative skin sensitization in Part A were assigned to Part B of the study. In Part B Participants received intradermal injections of EXC 001 on 1 side of the abdominal incisions and on the other side received intradermal injections of placebo matched to EXC 001 at Week 2, 4, 6, 8 and 10. On the EXC 001 treated side 1 column received high dose (5.0 mg/linear cm) and other a low dose (1.0 mg/linear cm). Out of 2 lateral biomarker incisions 1 incision received high dose (5.0 mg/linear cm) and other a low dose (1.0 mg/linear cm). Participants received an abdominoplasty at week 13 with a follow-up post-surgery visit at week 14.
- Cohort 2: EXC 001 and Placebo: In Part A participants received single intradermal injections of EXC-001 at a dose of 5 milligram (mg) on Day 1 and 21. Third 5 mg intradermal injection was administered at the discretion of Investigator based on the event of an equivocal skin sensitization on Day 38 or at least 7 days prior to surgery (Day 1 in Part B). The injection site was evaluated immediately after the injection and on Days 21, 28, 38, 50 until day of surgery. Participants with negative skin sensitization in Part A were assigned to Part B of the study. In Part B participants received intradermal injections of EXC 001 on 1 side of the abdominal incisions and on the other side received intradermal injections of placebo matched to EXC 001 at Week 2, 5, 8 and 11. On the EXC 001 treated side 1 column received high dose (5.0 mg/linear cm) and other a low dose (1.0 mg/linear cm). Out of 2 lateral biomarker incisions 1 incision received high dose (5.0 mg/linear cm) and other a low dose (1.0 mg/linear cm). Participants received an abdominoplasty at week 13 with a follow-up post-surgery visit at week 14.
- Cohort 3: EXC 001 and Placebo: In Part A participants received single intradermal injections of EXC-001 at a dose of 5 milligram (mg) on Day 1 and 21. Third 5 mg intradermal injection was administered at the discretion of Investigator based on the event of an equivocal skin sensitization on Day 38 or at least 7 days prior to surgery (Day 1 in Part B). The injection site was evaluated immediately after the injection and on Days 21, 28, 38, 50 until day of surgery. Participants with negative skin sensitization in Part A were assigned to Part B of the study. In Part B participants received intradermal injections of EXC 001 on 1 side of the abdominal incisions and on the other side received intradermal injections of placebo matched to EXC 001 at Week 2, 6 and 10. On the EXC 001 treated side 1 column received high dose (5.0 mg/linear cm) and other a low dose (1.0 mg/linear cm). Out of 2 lateral biomarker incisions 1 incision received high dose (5.0 mg/linear cm) and other a low dose (1.0 mg/linear cm). Participants received an abdominoplasty at week 13 with a follow-up post-surgery visit at week 14.
Period: Part A: Skin Testing Phase (50 Days)
Arm/Group | Cohort 1: EXC 001 and Placebo | Cohort 2: EXC 001 and Placebo | Cohort 3: EXC 001 and Placebo
Started | 10 | 10 | 10
Completed | 9 | 10 | 10
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Part B: Active Dosing Phase (13 Weeks)
Arm/Group | Cohort 1: EXC 001 and Placebo | Cohort 2: EXC 001 and Placebo | Cohort 3: EXC 001 and Placebo
Started | 9 | 10 | 10
Completed | 9 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included participants who completed Day 1 of Part A and received at least 1 dose of study drug.
Groups:
- Cohort 1: EXC 001 and Placebo: In Part A participants received single intradermal injections of EXC-001 at a dose of 5 mg on Day 1 and 21. Third 5 mg intradermal injection was administered at the discretion of Investigator based on the event of an equivocal skin sensitization on Day 38 or at least 7 days prior to surgery (Day 1 in Part B). The injection site was evaluated immediately after the injection and on Days 21, 28, 38, 50 until day of surgery. Participants with negative skin sensitization in Part A were assigned to Part B of the study. In Part B Participants received intradermal injections of EXC 001 on 1 side of the abdominal incisions and on the other side received intradermal injections of placebo matched to EXC 001 at Week 2, 4, 6, 8 and 10. On the EXC 001 treated side 1 column received high dose (5.0 mg/linear cm) and other a low dose (1.0 mg/linear cm). Out of 2 lateral biomarker incisions 1 incision received high dose (5.0 mg/linear cm) and other a low dose (1.0 mg/linear cm). Participants received an abdominoplasty at week 13 with a follow-up post-surgery visit at week 14.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: EXC 001 and Placebo | Cohort 2: EXC 001 and Placebo | Cohort 3: EXC 001 and Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 10 | 29
  Male | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part B: Expert Panel Scar Assessment Score
Description: Scar assessment by an expert panel was done on blinded photographs using 100 millimeter (mm) visual analog scale (VAS) where a score of 0 mm = best possible scar and a score of 100 mm = worst possible scar, where higher scores indicate worse condition. The difference was calculated for scars at Week 13 as EXC 001 score minus placebo score, thus a negative difference would indicate that the EXC 001-treated scars had lower scar severity. The score was defined as the within participant average difference between EXC 001- and Placebo-treated scars at Week 13.
Time Frame: Week 13 of Part B
Population: Completer population included all participants who missed not more than 1 dose of study drug, had the Week 13 assessment and non-missing data for VAS scar assessment score for at least one dose level.
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Part B: Cohort 1: EXC 001 High Dose (5.0 mg/Linear cm) + Placebo: Participants received intradermal injections of EXC 001 high dose (5.0 mg/linear cm) in 1 vertical column and 1 lateral biomarker incision on 1 side of the abdominal incisions and intradermal injections of placebo matched to EXC 001 on the other side at Week 2, 4, 6, 8 and 10.
- Part B: Cohort 1: EXC 001 Low Dose (1.0 mg/Linear cm) + Placebo: Participants received intradermal injections of EXC 001 low dose (1.0 mg/linear cm) in 1 vertical column and 1 lateral biomarker incision on 1 side of the abdominal incisions and intradermal injections of placebo matched to EXC 001 on the other side at Week 2, 4, 6, 8 and 10.
- Part B: Cohort 2: EXC 001 High Dose (5.0 mg/Linear cm) + Placebo: Participants received intradermal injections of EXC 001 high dose (5.0 mg/linear cm) in 1 vertical column and 1 lateral biomarker incision on 1 side of the abdominal incisions and intradermal injections of placebo matched to EXC 001 on the other side at Week 2, 5, 8 and 11.
- Part B: Cohort 2: EXC 001 Low Dose (1.0 mg/Linear cm) + Placebo: Participants received intradermal injections of EXC 001 low dose (1.0 mg/linear cm) in 1 vertical column and 1 lateral biomarker incision on 1 side of the abdominal incisions and intradermal injections of placebo matched to EXC 001 on the other side at Week 2, 5, 8 and 11.
- Part B: Cohort 3: EXC 001 High Dose (5.0 mg/Linear cm) + Placebo: Participants received intradermal injections of EXC 001 high dose (5.0 mg/linear cm) in 1 vertical column and 1 lateral biomarker incision on 1 side of the abdominal incisions and intradermal injections of placebo matched to EXC 001 on the other side at Week 2, 6 and 10.
- Part B: Cohort 3: EXC 001 Low Dose (1.0 mg/Linear cm) + Placebo: Participants received intradermal injections of EXC 001 low dose (1.0 mg/linear cm) in 1 vertical column and 1 lateral biomarker incision on 1 side of the abdominal incisions and intradermal injections of placebo matched to EXC 001 on the other side at Week 2, 6 and 10.
Arm/Group | Part B: Cohort 1: EXC 001 High Dose (5.0 mg/Linear cm) + Placebo | Part B: Cohort 1: EXC 001 Low Dose (1.0 mg/Linear cm) + Placebo | Part B: Cohort 2: EXC 001 High Dose (5.0 mg/Linear cm) + Placebo | Part B: Cohort 2: EXC 001 Low Dose (1.0 mg/Linear cm) + Placebo | Part B: Cohort 3: EXC 001 High Dose (5.0 mg/Linear cm) + Placebo | Part B: Cohort 3: EXC 001 Low Dose (1.0 mg/Linear cm) + Placebo
Number analyzed (Participants) | 8 | 8 | 10 | 10 | 10 | 10
millimeters | -3.16 (7.687) | 0.18 (7.154) | 1.45 (12.450) | 2.91 (9.778) | -4.78 (11.326) | -4.05 (8.934)

2. Secondary Outcome: Part B: Physician Observer Global Assessment Scar Score
Description: Physician observer global assessment of scar score was done using a valid published 10-point rating scale. Physicians rated severity of each scar on a scale of 1 = normal skin to 10 = worst scar imaginable. Each scar was given a single score and the differences in scores between the matched pairs of scars were calculated. There were 4 differences within each dose level that were averaged to create a single score for each participant at each dose level. The score was defined as the within participant average difference between EXC 001 and Placebo.
Time Frame: Week 13 of Part B
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B: Cohort 1: EXC 001 High Dose (5.0 mg/Linear cm) + Placebo | Part B: Cohort 1: EXC 001 Low Dose (1.0 mg/Linear cm) + Placebo | Part B: Cohort 2: EXC 001 High Dose (5.0 mg/Linear cm) + Placebo | Part B: Cohort 2: EXC 001 Low Dose (1.0 mg/Linear cm) + Placebo | Part B: Cohort 3: EXC 001 High Dose (5.0 mg/Linear cm) + Placebo | Part B: Cohort 3: EXC 001 Low Dose (1.0 mg/Linear cm) + Placebo
Number analyzed (Participants) | 8 | 8 | 10 | 10 | 10 | 10
units on a scale | -0.84 (1.362) | -0.44 (1.193) | -0.68 (1.448) | -0.05 (0.848) | -0.75 (1.965) | -0.70 (1.153)

3. Secondary Outcome: Part B: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Following vital sign parameters were assessed: diastolic blood pressure, systolic blood pressure, respiration rate, pulse rate, temperature and weight. Number of participants with clinically significant change in any vital sign parameter compared to Baseline were reported. Criteria for clinically significant change in any vital sign parameter compared to baseline was based on investigator's discretion.
Time Frame: Part B: Day 1 up to Week 14
Population: Safety population included participants who completed Part A Day 1 visit of and received at least 1 dose of study drug. Safety assessment was not planned separately for EXC 001 and placebo in Part B. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: EXC 001 and Placebo | Cohort 2: EXC 001 and Placebo | Cohort 3: EXC 001 and Placebo
Number analyzed (Participants) | 9 | 10 | 10
Participants | 0 | 0 | 0

4. Secondary Outcome: Part B: Number of Participants With Clinically Significant Changes in Physical Examination Findings
Description: Physical examination included the assessment of skin; head, ears, eyes, nose, and throat; respiratory; cardiovascular; abdomen; musculoskeletal; neurological; gastrointestinal; genitourinary; endocrine and lymph nodes. Criteria for clinically significant findings in physical examination was based on investigator's discretion.
Time Frame: Part B: Day 1 up to Week 14
Population: Safety population included participants who completed Part A Day 1 visit of Part A and received at least 1 dose of study drug. Safety assessment was not planned separately for EXC 001 and placebo in Part B. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: EXC 001 and Placebo | Cohort 2: EXC 001 and Placebo | Cohort 3: EXC 001 and Placebo
Number analyzed (Participants) | 9 | 10 | 10
Participants | 1 | 0 | 1

5. Secondary Outcome: Part B: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Findings
Description: Following parameters were analyzed for ECG abnormality: PR interval, QRS interval, QT interval, QT interval corrected using the Fridericia's correction (QTc), heart rate (HR). A standard, single 12-lead ECG was taken and results was classified as normal, having a clinically insignificant abnormality, or having a clinically significant abnormality. Number of participants with clinically significant abnormality in ECG compared to baseline were reported. Criteria for clinically significant abnormality in ECG compared to baseline was based on investigator's discretion.
Time Frame: Week 13 of Part B
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: EXC 001 and Placebo | Cohort 2: EXC 001 and Placebo | Cohort 3: EXC 001 and Placebo
Number analyzed (Participants) | 9 | 10 | 10
Participants | 0 | 0 | 0

6. Secondary Outcome: Part B: Number of Participants With Clinically Significant Abnormal Laboratory Findings
Description: Laboratory analysis included hematology, biochemistry and urinalysis. Hematology range: basophils (bas) 0-0.2, eosinophils (eos) 0-0.4, leukocytes (leu) 4-10.5, lymphocytes (lym) 0.7-4.5, neutrophils (neu) 1.8-7.8, platelet 140-415, monocytes (mon) 0.1-1 in 10^9 per liter; bas/leu 0-3, eos/leu 0-7, lym/leu 14-46, mon/leu 4-13, neu/leu and neu/leu 40-74 in percentage, erythrocytes 3.8-5.1 10^12/L, hematocrit 0.34-0.44 L/L, hemoglobin 115-150 gram per liter (g/L). Biochemistry range: creatine kinase 24-173, alkaline phosphatase 25-150, alanine aminotransferase (AT) and aspartate AT 0-40 in International units per liter; creatinine 50-88, urate 89-399, bilirubin 2-21 in micromole per liter, glucose 3.6-5.5, potassium 3.5-5.5, sodium 135-148, blood urea nitrogen 1.8-9.3 in millimole/L, albumin 35-55 g/L. Urinalysis parameters: pH (5-7.5), specific gravity (1.005-1.03). Participants with clinically significant abnormal change in any laboratory parameter compared to baseline were reported.
Time Frame: Part B: Day 1 up to Week 13
Population: Safety population included participants who completed Part A Day 1 visit and received at least 1 dose of study drug. Safety assessment was not planned separately for EXC 001 and placebo in Part B. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: EXC 001 and Placebo | Cohort 2: EXC 001 and Placebo | Cohort 3: EXC 001 and Placebo
Number analyzed (Participants) | 9 | 10 | 10
Participants | 0 | 0 | 0

7. Secondary Outcome: Part A and B: Number of Participants With Positive Skin Sensitivity Reaction
Description: The skin sensitivity reaction was assessed only at the skin sensitivity reaction testing sites. Erythematous, raised (indurated) and edematous reactions were considered as positive skin sensitivity reactions. The number of participants that experienced any positive skin sensitivity reactions were reported.
Time Frame: From Day 21 of Part A up to Week 2 of Part B
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: EXC 001 and Placebo | Cohort 2: EXC 001 and Placebo | Cohort 3: EXC 001 and Placebo
Number analyzed (Participants) | 9 | 10 | 10
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Safety population included participants who completed Part A Day 1 visit of and received at least 1 dose of study drug. Safety assessment was not planned separately for EXC 001 and placebo in Part B.
Groups:
- Part A: Cohort 1: EXC 001; Part A: Cohort 2: EXC 001; Part A: Cohort 3: EXC 001: Participants received single intradermal injections of EXC-001 at a dose of 5 milligram (mg) on Day 1 and 21. Third 5 mg intradermal injection was administered at the discretion of Investigator based on the event of an equivocal skin sensitization on Day 38 or at least 7 days prior to surgery (Day 1 in Part B). The injection site was evaluated immediately after the injection and on Days 21, 28, 38, 50 until day of surgery. Participants with negative skin sensitization in Part A were assigned to Part B of the study.
- Part B: Cohort 1: EXC 001 and Placebo: Participants received intradermal injections of EXC 001 on 1 side of the abdominal incisions and on the other side received intradermal injections of placebo matched to EXC 001 at Week 2, 4, 6, 8 and 10. On the EXC 001 treated side 1 column received high dose (5.0 mg/linear cm) and other a low dose (1.0 mg/linear cm). Out of 2 lateral biomarker incisions 1 incision received high dose (5.0 mg/linear cm) and other a low dose (1.0 mg/linear cm). Participants received an abdominoplasty at week 13 with a follow-up post-surgery visit at week 14.
- Part B: Cohort 2: EXC 001 and Placebo: Participants received intradermal injections of EXC 001 on 1 side of the abdominal incisions and on the other side received intradermal injections of placebo matched to EXC 001 at Week 2, 5, 8 and 11. On the EXC 001 treated side 1 column received high dose (5.0 mg/linear cm) and other a low dose (1.0 mg/linear cm). Out of 2 lateral biomarker incisions 1 incision received high dose (5.0 mg/linear cm) and other a low dose (1.0 mg/linear cm). Participants received an abdominoplasty at week 13 with a follow-up post-surgery visit at week 14.
- Part B: Cohort 3: EXC 001 and Placebo: Participants received intradermal injections of EXC 001 on 1 side of the abdominal incisions and on the other side received intradermal injections of placebo matched to EXC 001 at Week 2, 6 and 10. On the EXC 001 treated side 1 column received high dose (5.0 mg/linear cm) and other a low dose (1.0 mg/linear cm). Out of 2 lateral biomarker incisions 1 incision received high dose (5.0 mg/linear cm) and other a low dose (1.0 mg/linear cm). Participants received an abdominoplasty at week 13 with a follow-up post-surgery visit at week 14.
Arm/Group | Part A: Cohort 1: EXC 001 | Part A: Cohort 2: EXC 001 | Part A: Cohort 3: EXC 001 | Part B: Cohort 1: EXC 001 and Placebo | Part B: Cohort 2: EXC 001 and Placebo | Part B: Cohort 3: EXC 001 and Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/9 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 2/10 | 1/10 | 9/9 | 8/10 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Cohort 1: EXC 001 (N=10) | Part A: Cohort 2: EXC 001 (N=10) | Part A: Cohort 3: EXC 001 (N=10) | Part B: Cohort 1: EXC 001 and Placebo (N=9) | Part B: Cohort 2: EXC 001 and Placebo (N=10) | Part B: Cohort 3: EXC 001 and Placebo (N=10)
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 6 | 6 | 7
Incision site pruritus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 2
Incision site oedema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Incision site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.